CLINICAL TRIAL: NCT04250298
Title: Pilot Study to Gain First Indications for the Impact of a Three-month's Oral Intake of an Iron Supplement With High Bioavailability on the Hemoglobin Concentration in Iron Deficient Blood Donors
Brief Title: Sucrosom5al Iron Supplementation in Blood Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Johannes Kepler University of Linz (Other); Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-435 ex 18/19
Record Dates: First submitted 2020-01-21; First posted 2020-01-31 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Iron-deficiency
Keywords: blood donors; donor rejection; sucrosomial iron; dietary supplements
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — sucrosomial iron

STUDY DESIGN:
Intervention Model Description: This monocentric study (single cohort study design) is classified as a food study (application of the commercially available supplement OLEOvital® EISEN FORTE) in an interventional setting (study-related measures: additional blood tests and oral intake of OLEOvital® EISEN FORTE).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iron deficient blood donors (Other): Daily intake of 30 mg of sucrosomial iron during 90-120 days (male and female whole blood donors)
  Interventions: Dietary Supplement: sucrosomial iron

INTERVENTIONS:
Dietary Supplement: sucrosomial iron — oral intake of iron as sachets or capsules
  Other Names: OLEOvital(R) EISEN FORTE

SUMMARY:
The aim of this descriptive/explorative pilot study is to examine the effects of supplementing a sucrosomial iron preparation in whole blood donors with iron deficiency for three months.

DETAILED DESCRIPTION:
In this academic, monocentric interventional pilot study with one cohorte, otherwise healthy blood donors who have been rejected from blood donation due to low hemoglobin (females <12.5 g/dl, males <13.5 g/dl) and low ferritin levels (<30 ng/ml) receive an iron-containing dietary supplement (sucrosomial iron) for three months with a daily intake of 30 g iron.

Fifty donors will be included in the study. The study population will consist of two sub-groups (premenopausal women and postmenopausal women plus men).

Our aim is to

* gain first findings concerning the extent of the change primarily in hemoglobin and secondly in ferritin concentrations
* observe acceptance and tolerance after intake of the test product for several months
* create pilot data for a following randomized controlled study.

In addition, possible clinical symptoms associated with iron deficiency will be recorded by using appropriate questionnaires (Questionnaire on the assessment of health-related quality of life [WHOQOL-Bref], Fatigue assessment questionnaire [FAQ], questionnaire on psychic symptoms of insomnia [RIS] and Restless Legs Syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Deferral from donation because of low capillary hemoglobin (Hb) <12.5 g/dl (women) and Hb <13 g/dl;
* Otherwise eligibility for donation according to medical history;
* Ferritin at the time of deferral <30 ng/ml;
* Last whole blood donation >2 months prior to current hemoglobin level;
* Written informed consent;
* Venous Hb <12.5 g/dl (females) and <13.5 g/dl (men);

Exclusion Criteria:

* Lack of legal capacity or court-appointed representation;
* Known pregnancy;
* Lactation period;
* Chronic diarrhea or known inclination for diarrhea;
* Known or suspected fructose intolerance;
* iron supplementation during the last three months;
* continuous or expected blood loss (capillary oozing);
* hypermenorrhea;
* planned surgical intervention with relevant blood loss within the next 3-4 months (duration of study);
* application of another iron supplementation during the next 3-4 months;
* intended application of preparations for a systematic increase of red blood cell and hemoglobin concentration or production (e.g. erythropoietin preparations, packed red blood cells) for the duration of the study;
* parallel participation in another clinical trial with insurance coverage;
* foreseeable compliance issues;
* foreseeable unavailability for the time of the final examination;
* Incompatibility with any of the ingredients of the product;
* Anemia requiring acute therapy: Hb <8g/dl (as indication of an obligatory correction of the hemoglobin level to a clinically irrelevant or non-therapeutic value);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- [Background] Bialkowski W, Bryant BJ, Schlumpf KS, Wright DJ, Birch R, Kiss JE, D'Andrea P, Cable RG, Spencer BR, Vij V, Mast AE. The strategies to reduce iron deficiency in blood donors randomized trial: design, enrolment and early retention. Vox Sang. 2015 Feb;108(2):178-85. doi: 10.1111/vox.12210. Epub 2014 Dec 3. PMID 25469720
- [Background] Finch CA, Cook JD, Labbe RF, Culala M. Effect of blood donation on iron stores as evaluated by serum ferritin. Blood. 1977 Sep;50(3):441-7. PMID 884321
- [Background] Cable RG, Glynn SA, Kiss JE, Mast AE, Steele WR, Murphy EL, Wright DJ, Sacher RA, Gottschall JL, Vij V, Simon TL; NHLBI Retrovirus Epidemiology Donor Study-II. Iron deficiency in blood donors: analysis of enrollment data from the REDS-II Donor Iron Status Evaluation (RISE) study. Transfusion. 2011 Mar;51(3):511-22. doi: 10.1111/j.1537-2995.2010.02865.x. Epub 2010 Aug 30. PMID 20804527
- [Background] Rigas AS, Sorensen CJ, Pedersen OB, Petersen MS, Thorner LW, Kotze S, Sorensen E, Magnussen K, Rostgaard K, Erikstrup C, Ullum H. Predictors of iron levels in 14,737 Danish blood donors: results from the Danish Blood Donor Study. Transfusion. 2014 Mar;54(3 Pt 2):789-96. doi: 10.1111/trf.12518. Epub 2013 Dec 23. PMID 24372094
- [Background] Conrad ME, Crosby WH, Jacobs A, Kaltwasser JP, Nusbacher J. The Hippocratian principle of 'primum nil nocere' demands that the metabolic state of a donor should be normalized prior to a subsequent donation of blood or plasma. How much blood, relative to his body weight, can a donor give over a certain period, without a continuous deviation of iron metabolism in the direction of iron deficiency? Vox Sang. 1981 Nov-Dec;41(5-6):336-43. doi: 10.1111/j.1423-0410.1981.tb01059.x. No abstract available. PMID 7324448
- [Background] Bianco C, Brittenham G, Gilcher RO, Gordeuk VR, Kushner JP, Sayers M, Chambers L, Counts RB, Aylesworth C, Nemo G, Alving B. Maintaining iron balance in women blood donors of childbearing age: summary of a workshop. Transfusion. 2002 Jun;42(6):798-805. doi: 10.1046/j.1537-2995.2002.00103.x. No abstract available. PMID 12147035
- [Background] Cable RG, Brambilla D, Glynn SA, Kleinman S, Mast AE, Spencer BR, Stone M, Kiss JE; National Heart, Lung, and Blood Institute Recipient Epidemiology and Donor Evaluation Study-III (REDS-III). Effect of iron supplementation on iron stores and total body iron after whole blood donation. Transfusion. 2016 Aug;56(8):2005-12. doi: 10.1111/trf.13659. Epub 2016 May 27. PMID 27232535
- [Background] Kiss JE, Brambilla D, Glynn SA, Mast AE, Spencer BR, Stone M, Kleinman SH, Cable RG; National Heart, Lung, and Blood Institute (NHLBI) Recipient Epidemiology and Donor Evaluation Study-III (REDS-III). Oral iron supplementation after blood donation: a randomized clinical trial. JAMA. 2015 Feb 10;313(6):575-83. doi: 10.1001/jama.2015.119. PMID 25668261
- [Background] Moretti D, Goede JS, Zeder C, Jiskra M, Chatzinakou V, Tjalsma H, Melse-Boonstra A, Brittenham G, Swinkels DW, Zimmermann MB. Oral iron supplements increase hepcidin and decrease iron absorption from daily or twice-daily doses in iron-depleted young women. Blood. 2015 Oct 22;126(17):1981-9. doi: 10.1182/blood-2015-05-642223. Epub 2015 Aug 19. PMID 26289639
- [Background] Stoffel NU, Cercamondi CI, Brittenham G, Zeder C, Geurts-Moespot AJ, Swinkels DW, Moretti D, Zimmermann MB. Iron absorption from oral iron supplements given on consecutive versus alternate days and as single morning doses versus twice-daily split dosing in iron-depleted women: two open-label, randomised controlled trials. Lancet Haematol. 2017 Nov;4(11):e524-e533. doi: 10.1016/S2352-3026(17)30182-5. Epub 2017 Oct 9. PMID 29032957
- [Background] Pisani A, Riccio E, Sabbatini M, Andreucci M, Del Rio A, Visciano B. Effect of oral liposomal iron versus intravenous iron for treatment of iron deficiency anaemia in CKD patients: a randomized trial. Nephrol Dial Transplant. 2015 Apr;30(4):645-52. doi: 10.1093/ndt/gfu357. Epub 2014 Nov 13. PMID 25395392
- [Background] Parisi F, Berti C, Mando C, Martinelli A, Mazzali C, Cetin I. Effects of different regimens of iron prophylaxis on maternal iron status and pregnancy outcome: a randomized control trial. J Matern Fetal Neonatal Med. 2017 Aug;30(15):1787-1792. doi: 10.1080/14767058.2016.1224841. Epub 2016 Sep 2. PMID 27588568
- [Background] Spencer BR, Kleinman S, Wright DJ, Glynn SA, Rye DB, Kiss JE, Mast AE, Cable RG; REDS-II RISE Analysis Group. Restless legs syndrome, pica, and iron status in blood donors. Transfusion. 2013 Aug;53(8):1645-52. doi: 10.1111/trf.12260. Epub 2013 Jun 13. PMID 23763445
- [Background] Verdon F, Burnand B, Stubi CL, Bonard C, Graff M, Michaud A, Bischoff T, de Vevey M, Studer JP, Herzig L, Chapuis C, Tissot J, Pecoud A, Favrat B. Iron supplementation for unexplained fatigue in non-anaemic women: double blind randomised placebo controlled trial. BMJ. 2003 May 24;326(7399):1124. doi: 10.1136/bmj.326.7399.1124. PMID 12763985
- [Background] Brownlie T 4th, Utermohlen V, Hinton PS, Haas JD. Tissue iron deficiency without anemia impairs adaptation in endurance capacity after aerobic training in previously untrained women. Am J Clin Nutr. 2004 Mar;79(3):437-43. doi: 10.1093/ajcn/79.3.437. PMID 14985219
- [Background] Murray-Kolb LE, Beard JL. Iron treatment normalizes cognitive functioning in young women. Am J Clin Nutr. 2007 Mar;85(3):778-87. doi: 10.1093/ajcn/85.3.778. PMID 17344500
- [Background] Moeinvaziri M, Mansoori P, Holakooee K, Safaee Naraghi Z, Abbasi A. Iron status in diffuse telogen hair loss among women. Acta Dermatovenerol Croat. 2009;17(4):279-84. PMID 20021982
- [Background] Chansky MC, King MR, Bialkowski W, Bryant BJ, Kiss JE, D'Andrea P, Cable RG, Spencer BR, Mast AE. Qualitative assessment of pica experienced by frequent blood donors. Transfusion. 2017 Apr;57(4):946-951. doi: 10.1111/trf.13981. Epub 2017 Feb 5. PMID 28164344
- [Background] Allen RP, Picchietti D, Hening WA, Trenkwalder C, Walters AS, Montplaisi J; Restless Legs Syndrome Diagnosis and Epidemiology workshop at the National Institutes of Health; International Restless Legs Syndrome Study Group. Restless legs syndrome: diagnostic criteria, special considerations, and epidemiology. A report from the restless legs syndrome diagnosis and epidemiology workshop at the National Institutes of Health. Sleep Med. 2003 Mar;4(2):101-19. doi: 10.1016/s1389-9457(03)00010-8. PMID 14592341

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: The arm includes male and female whole blood donors who were deferred from blood donation.
Period: Overall Study
Arm/Group | Single Arm
Started | 50
Completed | 47
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Per protocol evaluation
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.81 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 47
Hemoglobin [Median (Inter-Quartile Range); unit: g/dl] | 12.0 [11.6 to 12.2]
Ferritin [Median (Inter-Quartile Range); unit: ng/ml] | 8.71 [6.8 to 11.77]

OUTCOME MEASURES:

1. Primary Outcome: Hb (g/dl) at E2
Description: hemoglobin level after iron supplementation at examination 2 (E2, after iron intake over 90-120 days)
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, post menopausal or male
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Single Arm
Number analyzed (Participants) | 47
g/dl | 13.07 (1.03)
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.031, t-test, 2 sided

2. Primary Outcome: Δ Hb (g/dl) (E2-E1)
Description: Change of hemoglobin between visit 1 (E1, baseline ) prior to iron substitution and examination 2 (E2, after 90-120 days) after iron substitution
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Single Arm
Number analyzed (Participants) | 47
g/dl | 1.08 (0.9)
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.267, t-test, 2 sided

3. Primary Outcome: Δ Hb (g/dl) (E2-E1) / 90 Days
Description: Change of hemoglobin between examination 1 (E1, baseline) prior to iron substitution and examination 2 (E2, after 90-120 days) after iron substitution interpolated to 90 days
Time Frame: 90 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Mean (Standard Error); unit: g/dl
Arm/Group | Single Arm
Number analyzed (Participants) | 47
g/dl | 0.99 (0.86)
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.228, t-test, 2 sided

4. Primary Outcome: Δ Hb (g/dl) (E2-E1)* Ratio
Description: Change of hemoglobin ratio of prescribed/taken iron supplementation/ 90 days (E1, baseline; E2, after 90-120 days) For practical reasons, the period between the first and the second examination and thus the duration of iron intake varied from 90 to 120 days. Therefore, as a result, all outcomes were standardized ot 90 days by interpolation
Time Frame: 90 days
Population: 23 premenopausal, female 24 postmenopausal, female or men
Measure: Median (Inter-Quartile Range); unit: g/dl
Arm/Group | Single Arm
Number analyzed (Participants) | 47
g/dl | 0.94 [0.3 to 1.63]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.267, t-test, 2 sided

5. Primary Outcome: Δ Response 1
Description: Change of Hb between examination 1 and examination 2 /90 days ≥1.0 g/dl [yes/no] --> The number of subjects in whom the Hb value improved by at least 1 g/dl between E1 (baseline) and E2 (after 90-120 days, following iron supplementation intake)
Time Frame: 90 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Participants | 19
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p > 0.999, Fisher Exact

6. Primary Outcome: Δ Response 2
Description: Change of Hb between examination 1 and examination 2 /90 days ≥1.5 g/dl [yes/no] --> The number of subjects in whom the Hb value improved by at least 1.5 g/dl between E1 (baseline) and E2 (after 90-120 days of iron supplementation intake)
Time Frame: 90 days
Population: 23 premenopausal female 24 postmenopausal, female, or male
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Participants | 12
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.318, Fisher Exact

7. Primary Outcome: Δ Response 3
Description: Change of Hb between examination 1 and examination 2 (E2)/90 days ≥2.0 g/dl [yes/no] --> The number of subjects in whom the Hb value improved by at least 2 g/dl between E1 (baseline) and E2 (after 90-120 days of iron supplementation intake)
Time Frame: 90 days
Population: 23 premenopausal, female 24 postmenopausal, female or male
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Participants | 5
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.348, Fisher Exact

8. Primary Outcome: Ferritin (ng/ml) at E2
Description: Ferritin level after iron supplementation at examination 2 (E2, 90-120 days after iron supplementation)
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Single Arm
Number analyzed (Participants) | 47
ng/ml | 16.54 (7.52)
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.548, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Δ Ferritin (ng/ml) (E2-E1)
Description: Change of Hemoglobin between examination 1 (E1, baseline) prior to iron substitution and examination 2 (E2, after 90-120 days) after iron substitution
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Single Arm
Number analyzed (Participants) | 47
ng/ml | 6.23 (6.59)
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.401, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Δ Ferritin (ng/ml) (E2-E1) / 90 Days
Description: Change of ferritin between examination 1 (E1, baseline ) to examination 2 (E2, after 90-120 days) interpolated to 90 days
Time Frame: 90 days
Population: 23 premenopausal women, 10 postmenopausal women and 14 men completed the study
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Single Arm
Number analyzed (Participants) | 47
ng/ml | 4.97 [1.23 to 8.83]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.506, Wilcoxon (Mann-Whitney)

11. Primary Outcome: Δ Ferritin (ng/ml) (E2-E1) * Ratio Capsule Intake / 90 Days
Description: Difference of ferritin values in ng/ml by comparing levels at baseline and 90-120 days after iron supplementation (interpolated to 90 days) A positive value for mean is considered an improvement.
Time Frame: 90 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Single Arm
Number analyzed (Participants) | 47
ng/ml | 5.74 (6.05)
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.506, Wilcoxon (Mann-Whitney)

12. Primary Outcome: Intake Evaluation
Description: Evaluation of the intake of sucrosomial iron [problem-free yes/no] --> The number of participants who reported problems with the intake of the iron sachets
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Participants
  problems with iron intake | 3
  no problems with iron intake | 44

13. Primary Outcome: Problems With Intake
Description: The number of participants with problems taking sucrosomial iron is listed, categorised according to their complaints.
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
participants
  initially mild sleeping problems | 1
  initially mild cough irritations | 1
  sachets were not easy to open | 1
  Uncertainty about whether the sachets had already been taken | 1

14. Primary Outcome: Recommendation
Description: Will use of sucrosomial iron for other blood donors be recommended [yes/no] --> The number refers to the number of participants who would recommend taking the product to others.
Time Frame: day 90-120
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Participants
  yes | 45
  no | 2

15. Primary Outcome: Renewed Intake
Description: Will sucrosomial iron will be taken again in the given case
Time Frame: day 90-120
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Participants
  yes | 47
  no | 0

16. Primary Outcome: Assumed Adverse Effects
Description: Assumed test product adverse effects
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Participants
  initially problems falling asleep | 1
  loose stools on occasion | 1
  pain in fingers and joints 2 weeks after starting the iron supplements | 1
  no adverse effects reported | 44

17. Primary Outcome: Quality of Life by World Health Organization Quality of Life Assessment (E2)
Description: Assessment of Scores at E2 after 90-120 days of iron intake. The WHOQOL-Bref includes 26 items with values of 1-5 addressing 4 domains (neg. phrased items are reversed for analysis.) Higher scores denote a higher quality of life, but there are no cut-off points above or below which quality of life could be evaluated as poor or good.
  Physical health: 7 items (4-20) Psychic health: 6 items (4-20) Social relationships: 3 items (4-20) Environment: 8 items (4-20) Score calculation: Domain and facet scores are scaled in a positive direction where higher scores denote higher quality of life (without adjusting to WHOQOL-100).
  Conversion to the final score (summarizing all 4 domains) was not performed (only the differences between E1 and E2 were of interest).
Time Frame: 14 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Units on a scale
  physical health | 18.4 [18.04 to 18.76]
  psychic health | 17.55 [17.17 to 17.94]
  social relationships | 17.73 [17.07 to 18.39]
  environment | 18.57 [18.22 to 18.93]
Statistical Analysis 1: Comparison: Single Arm; sub-population 1 vs. sub-population 2: Parametric and nonparametric univariate tests: t-test for independent samples, Mann-Whitney-U test, Fisher's exact test, chi-square homogeneity test; normal distribution check by Kolmogorov-Smirnov test with Lilliefors -significance correction, type I error = 10%). Estimate the true effect size: Two-sided 95% confidence intervals (depending on the nature of the data sets: parametric, non-parametric or Clopper-Pearson) are calculated for all parameters; Test type: Other — Mann-Whitney U test, Fisher Exact, Chi-Squared, Kolmogorv-Smirnow; p = 0.919, Wilcoxon (Mann-Whitney)

18. Primary Outcome: Δ Quality of Life by World Health Organization Quality of Life Assessment (E1-E2)
Description: Differences in the WHOQOL BREF categories between E1 (baseline) and E2 (after 90-120 days of iron intake).
  The WHOQOL-Bref includes 26 items with values of 1-5 addressing 4 domains (neg. phrased items are reversed for analysis.) Higher scores denote a higher quality of life, but there are no cut-off points above or below which quality of life could be evaluated as poor or good.
  Physical health: 7 items (4-20) Psychic health: 6 items (4-20) Social relationships: 3 items (4-20) Environment: 8 items (4-20) Score calculation: Domain and facet scores are scaled in a positive direction where higher scores denote higer qualitiy of life (without adjusting to WHOQOL-100).
  Conversion to the final score (summarizing all 4 domains) was not performed (only the differences between E1 and E2 were of interest).
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Units on a scale
  physical health | 0.99 [0.53 to 1.44]
  psychic health | 0.33 [0.03 to 0.64]
  social relationships | 0.03 [-0.58 to 0.64]
  environment | 0.33 [0.11 to 0.55]

19. Primary Outcome: Fatigue Assessment Questionnaire (E2)
Description: Assessment of the score at E2 (after 90-120 days of iron intake). The Fatigue Assessment Questionnaire (FAQ) is a 20-item self-report scale evaluating symptoms of chronic fatigue. Values range from 0-3. The total score ranges from 0 to 60, with a higher score indicating more severe fatigue.
  The answers to the questions had to refer to the past week in accordance with the FAQ guidelines, so 7 days was given as the outcome measure time frame.
  The mean with confidence interval (95%) for fatigue at E2 is shown here.
Time Frame: 7 days
Population: 23 female premenopausal 24 female postmenopausal or male
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Units on a scale | 9.11 [6.47 to 11.76]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.033, t-test, 2 sided

20. Primary Outcome: Δ Fatigue Assessment Questionnaire (E1-E2)
Description: In the Fatigue Assessment Questionnaire (FAQ) fatigue was determined at E1 and E2. The Fatigue Assessment Questionnaire (FAQ) is a 20-item self-report scale evaluating symptoms of chronic fatigue. Values range from 0-3. The total score ranges from 0 to 60, with a higher score indicating more severe fatigue. In this outcome the change of fatigue between examination 1 (E1, baseline) and examination 2 (after 90-120 days of iron intake) was determined.
  The answers to the questions had to refer to the past week in accordance with the FAQ guidelines, so 7 days was given as the outcome measure time frame.
  The number of subjects with fatigue before and after the intervention was analysed. A reduction in the number is considered an improvement.
  The mean (difference) with confidence interval (95%) for fatigue (E1-E2) is shown here.
Time Frame: 7 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Units on a scale | -15.53 [-20.08 to -10.98]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.585, t-test, 2 sided

21. Primary Outcome: Regensburg Insomnia Scale at E2
Description: Symptoms of insomnia were determined at examination 2 after 90-120 days of iron intake. The questionnaire consists of 10 items with values of 0-4. Total scores range from 0 to 40 points with higher scores indicative of more psychophysiological insomnia. Scores from 0-12 are considered normal and scores above the cutoff (13+) are an indication of symptoms associated with insomnia.
  The questions in the questionnaire relate to the last 4 weeks, so the time of the results measurement was set at 28 days.
  The mean with confidence interval (95%) for insomnia at E2 is shown here.
Time Frame: 28 days
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Units on a scale | 7.39 [6.16 to 8.62]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.676, t-test, 2 sided

22. Primary Outcome: Δ Regensburg Insomnia Scale (E1-E2)
Description: Change of symptoms of insomnia between examination 1 and examination 2. Symptoms of insomnia (Regensburg Insomnia Scale) were determined at examination 1 and 2. In this outcome the difference between E1 (baseline) and E2 (after 90-120 days of iron intake) was determined.
  The questionnaire consists of 10 items with values of 0-4. Total scores range from 0 to 40 points with higher scores indicative of more psychophysiological insomnia. Scores from 0-12 are considered normal and scores above the cutoff (13+) are an indication of symptoms associated with insomnia. A reduction in the score between E1 and E2 is considered an improvement in sleep.
  The mean (difference) with confidence interval (95%) for insomnia (E1-E2) is shown here.
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Units on a scale | -1.35 [-2.31 to -0.39]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.314, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Restless Legs Syndrome at E1
Description: The number of participants suffering from restless legs syndrome at baseline (E1)
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Count of Participants; unit: Participants
Groups:
- Iron Deficient Blood Donors: The arm includes male and female whole blood donors who were deferred from blood donation.
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
Participants | 6

24. Secondary Outcome: Restless Legs Syndrome at E2
Description: The number of participants suffering from restless legs syndrome at baseline (E2)
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or male
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
Participants | 3

25. Secondary Outcome: Frequency of Diarrhoea During Sucrosomial Iron Intake [Days]
Description: The number of participants who experienced diarrhoea during iron intake in days
Time Frame: 90-120 days
Population: 23 female premenopausal 24 female post menopausal or male
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
Participants | 0

26. Secondary Outcome: Clinical Symptoms of Iron Deficiency E1
Description: Clinical symptoms of iron deficiency at baseline (E1), numbers discribe the count of participants affected.
Time Frame: 90-120 days
Population: 23 female premenopausal 24 female post menopausal or male
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
participants
  brittle nails | 17
  increased hair loss | 13
  load dependant headache | 5
  shortness of breath | 13
  dizzyness | 7
  painful or "smooth" tongue | 1
  inexplicable food cravings | 0

27. Other Pre Specified Outcome: Hb at E1
Description: Hemoglobin at examination 1 (E1, baseline)
Time Frame: day 1
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
g/dl | 11.99 (0.59)
Statistical Analysis 1: Comparison: Iron Deficient Blood Donors; Test type: Other; p = 0.031, t-test, 2 sided

28. Other Pre Specified Outcome: Regensburg Insomnia Scale at E1
Description: Symptoms of insomnia at examination 1 (E1, baseline) Symptoms of insomnia were determined at E 1 prior iron intake (baseline). The questionnaire consists of 10 items with values of 0-4. Total scores range from 0 to 40 points with higher scores indicative of more psychophysiological insomnia. Scores from 0-12 are considered normal and scores above the cutoff (13+) are an indication of symptoms associated with insomnia.
  The questions in the questionnaire relate to the last 4 weeks, so the time of the results measurement was set at 28 days.
  The mean with confidence interval (95%) for insomnia at E1 is shown here.
Time Frame: 28 days
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
Units on a scale | 8.96 [7.49 to 10.42]
Statistical Analysis 1: Comparison: Iron Deficient Blood Donors; Test type: Other; p = 0.862, t-test, 2 sided

29. Other Pre Specified Outcome: RLS at E1
Description: Restless legs syndrome at examination 1 (E1, baseline) [yes/no]
Time Frame: day 1
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
Participants
  yes | 6
  no | 41
Statistical Analysis 1: Comparison: Iron Deficient Blood Donors; Test type: Other; p = 0.250, Fisher Exact

30. Other Pre Specified Outcome: Age at E1
Description: Age at examination 1 (E1, baseline) [years]
Time Frame: day 1
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
years | 42.81 (12.88)
Statistical Analysis 1: Comparison: Iron Deficient Blood Donors; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)

31. Other Pre Specified Outcome: Sex
Description: Sex [female/male]
Time Frame: day 1
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
Participants
  male | 14
  female, premenopausal | 23
  female,postmenopausal | 10
Statistical Analysis 1: Comparison: Iron Deficient Blood Donors; Test type: Other; p = 0.001, Fisher Exact

32. Other Pre Specified Outcome: Body Weight
Description: Body weight at examination 1 (E1, baseline) [kg]
Time Frame: day 1
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
kg | 69.45 (14.82)
Statistical Analysis 1: Comparison: Iron Deficient Blood Donors; Test type: Other; p = 0.055, Wilcoxon (Mann-Whitney)

33. Other Pre Specified Outcome: Body Heights
Description: Body heights at examination 1 (E1, baseline) [cm]
Time Frame: day 1
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
cm | 169.68 (9.15)
Statistical Analysis 1: Comparison: Iron Deficient Blood Donors; Test type: Other; p = 0.111, Wilcoxon (Mann-Whitney)

34. Other Pre Specified Outcome: BMI
Description: Body mass index at examination 1 (E1, baseline)
Time Frame: day 1
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
kg/m2 | 24.01 (3.92)
Statistical Analysis 1: Comparison: Iron Deficient Blood Donors; Test type: Other; p = 0.100, Wilcoxon (Mann-Whitney)

35. Other Pre Specified Outcome: Intake of Sucrosomial Iron I
Description: Participants could choose between sachets or capsules
Time Frame: day 1
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
Participants
  sachets | 47
  capsules | 0

36. Other Pre Specified Outcome: Intake Number
Description: Number of sachets or capsules (one per day) taken at E2 (after 90-120 days) [number]
Time Frame: day 90-120
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (Standard Deviation); unit: capsules/sachets
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
capsules/sachets | 98.13 (8.19)

37. Other Pre Specified Outcome: Intake Ratio
Description: Ratio of ingested to prescribed capsules
Time Frame: day 90-120
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
ratio | 1.03 (0.04)
Statistical Analysis 1: Comparison: Iron Deficient Blood Donors; Test type: Other; p = 0.111, Wilcoxon (Mann-Whitney)

38. Other Pre Specified Outcome: No Intake
Description: days of violation of the intake rules [days], where iron was not taken during the study interval
Time Frame: day 90-120
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
days | 2.77 (3.75)
Statistical Analysis 1: Comparison: Iron Deficient Blood Donors; Test type: Other; p = 0.213, Wilcoxon (Mann-Whitney)

39. Other Pre Specified Outcome: Number of Participants Who Met Drop Out Criteria
Description: Drop out criteria [categories] occuring during the study interval (between E1 and E2)
Time Frame: between E1 and E2
Population: 25 female, premenopausal 25 female, postmenopausal or men
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 50
Participants | 3

40. Other Pre Specified Outcome: Relevant Pre-existing Conditions
Description: relevant already cured pre-existing conditions [categories by type] prior to study begin
Time Frame: day 1
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
Participants | 0

41. Other Pre Specified Outcome: SAE
Description: Serious adverse events [categories by dype and duration]
Time Frame: 90-120 days
Population: 23 female, premenopausal 24 female, postmenopausal or men
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 47
Participants | 0

42. Other Pre Specified Outcome: Last Menstrual Period I
Description: Time interval between the end of the last menstrual period and blood collection for examination 1 (baseline) [days]
Time Frame: 0-90 days
Population: 23 premenopausal, female
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 23
days | 17.74 (10.32)

43. Other Pre Specified Outcome: Last Menstrual Period II
Description: Time interval between the end of the last menstrual period up to examination 2 (end of study interval after iron intake) [days]
Time Frame: 90-120 days
Population: 23 female, premenopausal
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 23
days | 16.48 (8.99)

44. Other Pre Specified Outcome: Last Menstrual Period III
Description: Count of menstrual bleedings between blood tests (during study interval) [number]
Time Frame: 90-120 days
Population: 23 premenopausal, female
Measure: Mean (Standard Deviation); unit: counts
Arm/Group | Iron Deficient Blood Donors
Number analyzed (Participants) | 23
counts | 2.91 (1.02)

45. Secondary Outcome: Clinical Symptoms of Iron Deficiency E2
Description: Clinical symptoms of iron deficiency at baseline (E2), numbers discribe the count of participants affected.
Time Frame: 90-120 days
Population: 23 female premenopausal 24 female post menopausal or male
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 47
participants
  brittle nails | 11
  increased hair loss | 8
  load dependant headache | 6
  shortness of breath | 9
  dizzyness | 6
  painful or "smooth" tongue | 0
  inexplicable food cravings | 1

ADVERSE EVENTS:
Time Frame: Adverse events were queried at the second visit, i.e. 90-120 days after the first visit.
Description: We used a food supplement in the dosage recommended by the manufacturer, already known to be well tolerated in (apart from iron deficiency) healthy blood donors. Therefore neither serious adverse events, nor a risk for all-cause mortality was expected.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 3/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=47)
Sleep (General disorders) | 1 (1) — initially problems to fall asleep
stool (Gastrointestinal disorders) | 1 (1) — occasionally loose stools
pain (General disorders) | 1 (1) — pain in fingers and wrists 2 weeks after start of iron supplementation

LIMITATIONS AND CAVEATS:
Single arm study without control group; small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT04250298/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT04250298/ICF_001.pdf